CLINICAL TRIAL: NCT00284557
Title: Evaluation of a Primary Care-Based Behavioral Intervention for Improving Physical Activity and Nutrition Behaviors Among High-Risk African-American Youth
Brief Title: A Primary Care Behavioral Approach for Addressing Childhood Overweight
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Anne Lang Dunlop, MD, MPH, Asst Professor, Emory University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 416-2005
Record Dates: First submitted 2006-01-30; First posted 2006-02-01 (Estimated); Results first posted 2012-06-28 (Estimated); Last update posted 2012-07-11 (Estimated); Status verified 2012-06

CONDITIONS: Obesity
Keywords: Behavioral/Social; Obesity; Pediatrics; Preventive Medicine
MeSH Terms: conditions — Obesity; Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group-based behavioral intervention (Experimental): The group-based behavioral intervention targets eating behaviors, physical activity, and "screen time", and is delivered to participating children and their parent/caregiver over the course of 4 weeks. Maintenance sessions occur every 3 months thereafter.
  Interventions: Behavioral: Group-based behavioral intervention
- Health education materials only (Active Comparator): Those allocated to Group 2 were provided with a standardized packet of health education materials addressing the recommended items from the expert committee guidelines (e.g., dietary recommendations using the Food Guide Pyramid and the Traffic Light Diet, a general prescription to increase physical activity to 60 minutes daily). They were also given a community resource list that provides contact and program information for community-based obesity treatment activities in their area.
  Interventions: Behavioral: Group-based behavioral intervention

INTERVENTIONS:
Behavioral: Group-based behavioral intervention — The group-based behavioral intervention targets eating behaviors, physical activity, and "screen time", and is delivered to participating children and their parent/caregiver over the course of 4 weeks. Maintenance sessions occur every 3 months thereafter.

SUMMARY:
The purpose of this study is to determine whether participation in a group-based health education curriculum is superior to receipt of standardized health educational materials for children who are overweight or at risk for overweight with regard to achievement of a healthier body weight and improvement of key eating and physical activity behaviors.

DETAILED DESCRIPTION:
In the United States, childhood obesity has tripled since 1970 such that 15% of those 6 to 19 years of age are obese, with higher observed prevalences for African-American and Hispanic children. Childhood obesity has significant short- and long-term health consequences. To avoid future morbidity, children who are obese or at risk for obesity must be identified and treated at an early stage. The primary care setting, where most children receive health care and where BMI should be tracked, may represent an early opportunity for identifying and treating childhood obesity. However, translational research is needed to test whether existing strategies for childhood obesity can be adapted for delivery via the primary care setting

The ultimate purpose of this work is to help overweight children, particularly those who are African-American, optimize their lifespan and quality of health through achievement of a healthier body mass index (BMI). Specific aims are to perform outcome and process evaluations to determine whether the intervention results in improvement in BMI percentile or habitual healthy eating and physical activity behaviors, and whether the intervention is feasible. The outcome evaluation component involves a randomized controlled trial, in which overweight children (BMI for age percentile >=95th) and children at risk for overweight (BMI for age percentile 85-94th)together with a parent/caregiver receive the primary care-based intervention or health education materials only. The intervention will focus on four main behavioral changes: decreasing consumption of key calorie-dense foods, increasing consumption of fruits and vegetables to ≥ 5 a day, reducing targeted sedentary behaviors to < 15 hrs per week, and increasing moderate and vigorous physical activity to 60 minutes or more daily. We will assess change in BMI percentile, number of servings of calorie-dense foods daily, and percent of time spent in sedentary and physical activities at 6-, 12-, and 18-months using mixed-model ANCOVA for repeated measures.

ELIGIBILITY:
Inclusion criteria included that the child must be:

1. Obese (BMI ≥ 95th percentile for age and gender) or at-risk for obesity (85th ≥ BMI > 95th percentile for age and gender);
2. African-American by parent report;
3. 7-11 years of age;
4. Without any medical or psychological condition that would make weight loss or physical activity dangerous, or psychological disorders that would make adoption of health behaviors difficult;
5. Without any complications of obesity that indicate prompt referral to a pediatric obesity treatment center for more aggressive weight loss therapy;
6. Together with the parent/caregiver indicate that they are ready to make changes in their eating and physical activity behaviors;
7. Have a parent/caregiver willing to participate.

Exclusion Criteria:

As noted above, to participate in this study the child must not have a medical or psychological condition that would make weight loss or physical activity dangerous, psychological disorders that would make adoption of health behaviors difficult, or complications of obesity that necessitate prompt referral to a pediatric obesity treatment center for more aggressive weight loss therapy. Examples of medical or psychological conditions that would render the child ineligible for this study include uncontrolled or poorly-controlled asthma or hypertension, bulimia, mental retardation or severe learning disability, as well as pseudotumor cerebri, sleep apnea, obesity hypoventilation syndrome, and slipped capital femoral epiphysis.

Ages: 7 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 130 (Actual)
Dates: Start 2006-01; Primary Completion 2010-03 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anne L Dunlop, MD, MPH, Principal Investigator — Emory University

RESULTS

PARTICIPANT FLOW:
Groups:
- Health Education Materials Only: Parent-child dyads allocated to Group 2 were provided with a standardized packet of health education materials addressing the recommended items from the expert committee guidelines (e.g., dietary recommendations using the Food Guide Pyramid and the Traffic Light Diet, a general prescription to increase physical activity to 60 minutes daily). They were also given a community resource list that provides contact and program information for community-based obesity treatment activities in their area.
Period: Overall Study
Arm/Group | Group-based Behavioral Intervention | Health Education Materials Only
Started | 67 | 63
Completed | 58 | 50
Not Completed | 9 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group-based Behavioral Intervention | Health Education Materials Only | Total
Number analyzed (Participants) | 67 | 63 | 130
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 67 | 63 | 130
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 9.5 (1.7) | 9.3 (1.4) | 9.4 (1.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49 | 45 | 94
  Male | 18 | 18 | 36
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 67 | 63 | 130
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 67 | 63 | 130

OUTCOME MEASURES:

1. Primary Outcome: BMI Z-score(for Gender and Age)at 6-months
Description: The body mass index (BMI) for a given age (in years and monthys) and gender (male or female) converted to an exact z-score.
Time Frame: 6-months post-intervention
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Group-based Behavioral Intervention | Health Education Materials Only
Number analyzed (Participants) | 61 | 54
Z-score | -0.129 (0.21) | 0.001 (0.16)

2. Secondary Outcome: Change in Eating Behaviors (Consumption of WHOA Foods), Physical Activity, and "Screen Time"
Time Frame: 6- and 12-months post-intervention
Reporting Status: Not Posted

3. Primary Outcome: BMI Z-score(for Gender and Age)at 12-months
Description: as for outcome 1
Time Frame: 12-months post-intervention
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Group-based Behavioral Intervention | Health Education Materials Only
Number analyzed (Participants) | 58 | 50
Z-score | -0.090 (0.29) | 0.001 (0.18)

ADVERSE EVENTS:
Arm/Group | Group-based Behavioral Intervention | Health Education Materials Only
Serious Adverse Events (participants affected / at risk) | 0/67 | 0/63
Other Adverse Events (participants affected / at risk) | 0/67 | 0/63

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes